CLINICAL TRIAL: NCT04340843
Title: A Phase 2 Study of Belinostat and SGI-110 (Guadecitabine) or ASTX727 for the Treatment of Unresectable and Metastatic Conventional Chondrosarcoma
Brief Title: Testing the Combination of Belinostat and SGI-110 (Guadecitabine) or ASTX727 for the Treatment of Unresectable and Metastatic Conventional Chondrosarcoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2020-02187; NCI-2020-02187 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10330 (Other: Yale University Cancer Center LAO); 10330 (Other: CTEP); UM1CA186686 (NIH)
Record Dates: First submitted 2020-04-09; First posted 2020-04-10 (Actual); Results first posted 2025-09-16 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Locally Advanced Unresectable Primary Central Chondrosarcoma; Metastatic Primary Central Chondrosarcoma; Unresectable Primary Central Chondrosarcoma
MeSH Terms: interventions — belinostat; Biopsy; Specimen Handling; decitabine and cedazuridine drug combination; guadecitabine; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (belinostat, guadecitabine, ASTX727) (Experimental): Patients receive guadecitabine SC or ASTX727 PO on days 1-5. Patients also receive belinostat IV over 30 minutes on days 1-5. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo collection of blood during screening, tumor biopsy during screening and on study, and MRI or CT throughout the trial.
  Interventions: Drug: Belinostat; Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Decitabine and Cedazuridine; Drug: Guadecitabine; Procedure: Magnetic Resonance Imaging

INTERVENTIONS:
Drug: Belinostat — Given IV
  Other Names: Beleodaq; PXD 101; PXD-101; PXD101
Procedure: Biopsy Procedure — Undergo biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo collection of blood
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Drug: Decitabine and Cedazuridine — Given PO
  Other Names: ASTX 727; ASTX-727; ASTX727; C-DEC; CDA Inhibitor E7727/Decitabine Combination Agent ASTX727; Cedazuridine/Decitabine Combination Agent ASTX727; Cedazuridine/Decitabine Tablet; DEC-C; Inaqovi; Inqovi
Drug: Guadecitabine — Given SC
  Other Names: DNMT inhibitor SGI-110; S110; SGI 110; SGI-110; SGI110
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI

SUMMARY:
This phase II trial studies the effect of belinostat and SGI-110 (guadecitabine) or ASTX727 in treating patients with conventional chondrosarcoma that cannot be removed by surgery (unresectable) and has spread from where it first started (primary site) to other places in the body (metastatic). Belinostat may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Chemotherapy drugs, such as guadecitabine and ASTX727, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving belinostat in combination with guadecitabine or ASTX727 may lower the chance of unresectable and metastatic chondrosarcoma growing or spreading.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To conduct a phase 2 clinical trial to evaluate whether combination treatment with belinostat and decitabine and cedazuridine (ASTX727) shows preliminary evidence of clinical activity in unresectable or metastatic conventional chondrosarcoma (CS) using an objective response rate endpoint.

SECONDARY OBJECTIVES:

I. To evaluate the toxicity profile associated with the belinostat and ASTX727. II. To evaluate the progression free survival (PFS) associated with the belinostat and ASTX727.

III. To evaluate the toxicity profile, objective response rate and progression free survival among the initial six patients treated with belinostat and SGI-110 (guadecitabine) prior to Amendment 5 in which ASTX727 was substituted for SGI-110 (guadecitabine).

CORRELATIVE OBJECTIVES:

I. To determine the IDH1/2 mutational status of subject's tumors and to evaluate for a relationship between presence of IDH1/2 mutation and clinical benefit from study treatment.

II. To conduct ribonucleic acid sequencing (RNAseq) analysis using baseline and on-treatment tissue biopsies to study the effects of study treatment on CS gene expression patterns and identify candidate genes which may underlie treatment efficacy.

III. To evaluate for changes in global deoxyribonucleic acid (DNA) methylation levels using baseline and on-treatment biopsies and correlate changes in global methylation with clinical benefit from study treatment.

IV. To use multiplex immunohistochemistry to interrogate the immune microenvironment in baseline and on-treatment tissue biopsies to define changes in infiltrating immune cell subsets and PD-L1/major histocompatibility complex (MHC) expression by immune and tumor cells associated with study treatment.

OUTLINE:

Patients receive guadecitabine subcutaneously (SC) or ASTX727 orally (PO) on days 1-5. Patients also receive belinostat intravenously (IV) over 30 minutes on days 1-5. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo collection of blood during screening, tumor biopsy during screening and on study, and magnetic resonance imaging (MRI) or computed tomography (CT) throughout the trial.

After completion of study treatment, patients are followed up every 3 months for 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have biopsy-proven conventional chondrosarcoma (CS) which is:

  * Either metastatic or locally advanced and unresectable, and
  * Measurable at study entry according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 criteria, and
  * Amenable to biopsy with imaging guidance at no or acceptable risk to the patient as defined by institutional guidelines for research-related biopsies or the treating investigator's assessment
  * In addition, the following criteria must be met:

    * Patients must have at least one lesion measurable by RECIST version 1.1 criteria which has not been previously irradiated
    * Patients who have histologic evidence of grade 1 chondrosarcoma only must either be symptomatic from their disease in the opinion of the treating investigator or demonstrate radiographic evidence of disease progression in the 3 months prior to initiation of study treatment
  * Note: Pathology review and confirmation of diagnosis will occur at the site enrolling the patient on this study
* Patients may have been treated with any number of prior systemic therapies. Because there are no Food and Drug Administration (FDA)-approved treatments for this disease, patients who have received no prior systemic therapy are also eligible. However, disease must be deemed surgically unresectable
* Age >= 18 years. Chondrosarcoma is rarely encountered in children and adolescents
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Absolute neutrophil count >= 1,000/mm^3
* Hemoglobin 8 g/dL
* Platelet count >= 75,000/mm^3
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2 x institutional ULN
* Creatinine =< 1.5 x institutional ULN OR glomerular filtration rate (GFR) >= 45 mL/min/1.73 m^2
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression, if patients have been clinically asymptomatic, and if patients have not received systemic corticosteroids for at least 28 days. Patients with brain metastases not meeting these criteria are not eligible
* Patients must be disease-free of prior invasive malignancies for > 5 years, with the exception of curatively-treated basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix.

  * NOTE: If there is a history of prior malignancy, patients must not be receiving other specific treatment for that cancer
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better
* The effects of belinostat and SGI-110 (guadecitabine) or ASTX727 on the developing human fetus are unknown. For this reason, and because the DNA methyltransferase inhibitor decitabine, the active metabolite of SGI-110 (guadecitabine) and a component of ASTX727, is known to be teratogenic, and because belinostat may cause teratogenicity and/or embryo-fetal lethality by virtue of targeting actively dividing cells, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation and for at least 6 months after the last dose of study drugs. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 3 months after completion of belinostat and SGI-110 (guadecitabine) or ASTX727 administration
* Patients must be able to understand and willing to sign a written informed consent document. Participants with impaired decision-making capacity (IDMC) who have a legally-authorized representative (LAR) and/or family member available will also be eligible

Exclusion Criteria:

* Patients with dedifferentiated, mesenchymal, or clear cell chondrosarcoma are not eligible
* Patients who have not recovered from adverse events (AEs) (i.e., have residual toxicities > grade 1) due to prior anti-cancer therapy are not allowed, with the exceptions of alopecia and endocrinopathies from prior immunotherapy-based treatments that are well-controlled with hormone replacement. In addition, the following time periods must elapse between the last dose of prior anti-cancer treatment and initiation of study treatment on this protocol:

  * Cytotoxic chemotherapy or biologic, including immunotherapy: 28 days
  * Small molecule targeted drug: 21 days or 5 half-lives, whichever is shorter. If 5 half-lives is shorter than 21 days, then 21 days applies.
  * Radiation: 28 days, except for palliative radiation, for which 14 days applies
* Patients who are receiving any other investigational agents
* Patients with known history of allergic reactions or sensitivity attributed to compounds of similar chemical or biologic composition to SGI-110 (guadecitabine), its active metabolite decitabine, or ASTX727, or belinostat
* Chronic use of any medications or substances that are strong inhibitors of UGT1A1 is not allowed. Patients must switch to alternative medications 7-14 days before treatment with belinostat. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated medical reference. As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product
* Patients with any known UGT1A1 polymorphism, heterozygous or homozygous, associated with reduced function (UGT1A1*6, UGT1A1*28, or UGT1A1*60)
* Patients with uncontrolled intercurrent illness
* Patients with psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because SGI-110 (guadecitabine) is a derivative of decitabine, and ASTX727 contains the agent decitabine, which has the potential for teratogenic or abortifacient effects, and because belinostat may cause teratogenicity and/or embryo-fetal lethality by virtue of targeting actively dividing cells. Because there is an unknown but potential risk for AEs in nursing infants secondary to treatment of the mother with SGI-110 (guadecitabine), ASTX727 and belinostat, breastfeeding should be discontinued
* Prolongation of the heart-rate corrected QT (QTc) interval >= 450 ms (i.e., grade 1 or higher) on the screening electrocardiogram (ECG) prior to initiation of study treatment. If baseline QTc on screening ECG is >= 450 ms (i.e., grade 1 or higher):

  * Check potassium and magnesium serum levels, and
  * Correct any identified hypokalemia and/or hypomagnesemia and repeat ECG to confirm a QTc interval < 450 ms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2020-09-08 (Actual); Primary Completion 2024-02-22 (Actual); Study Completion 2026-06-17 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Mia Weiss, Principal Investigator — Yale University Cancer Center LAO
Locations (39):
- United States (39):
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - USC Norris Oncology/Hematology-Newport Beach, Newport Beach, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Yale University, New Haven, Connecticut
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Northwestern University, Chicago, Illinois
  - HaysMed, Hays, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Mercy Hospital Pittsburg, Pittsburg, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - University Health Truman Medical Center, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - University of Kansas Cancer Center at North Kansas City Hospital, North Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - M D Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm

REFERENCES:
- [Derived] Sheikh TN, Chen X, Xu X, McGuire JT, Ingham M, Lu C, Schwartz GK. Growth Inhibition and Induction of Innate Immune Signaling of Chondrosarcomas with Epigenetic Inhibitors. Mol Cancer Ther. 2021 Dec;20(12):2362-2371. doi: 10.1158/1535-7163.MCT-21-0066. Epub 2021 Sep 22. PMID 34552007

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Belinostat, SGI-110): Patients receive SGI-110 (guadecitabine) SC on days 1-5. Patients also receive belinostat IV over 30 minutes on days 1-5. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo collection of blood during screening, tumor biopsy during screening and on study, and MRI or CT throughout the trial.
- Treatment (Belinostat, ASTX727): Patients receive ASTX727 (decitabine/cedazuridine) PO on days 1-5. Patients also receive belinostat IV over 30 minutes on days 1-5. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo collection of blood during screening, tumor biopsy during screening and on study, and MRI or CT throughout the trial.
Period: Overall Study
Arm/Group | Treatment (Belinostat, SGI-110) | Treatment (Belinostat, ASTX727)
Started | 6 | 13
Completed | 6 | 9
Not Completed | 0 | 4
Not completed — Adverse Event | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Treatment (Belinostat, ASTX727): Patients receive ASTX727 ((decitabine/cedazuridine) PO on days 1-5. Patients also receive belinostat IV over 30 minutes on days 1-5. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo collection of blood during screening, tumor biopsy during screening and on study, and MRI or CT throughout the trial.
- Total: Total of all reporting groups
Arm/Group | Treatment (Belinostat, SGI-110) | Treatment (Belinostat, ASTX727) | Total
Number analyzed (Participants) | 6 | 13 | 19
Age, Customized [Median (Full Range); unit: years]
  Age | 49.5 [42 to 62] | 67 [21 to 86] | 62 [21 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 4 | 10 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 5 | 12 | 17
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 1 | 2
  White | 5 | 12 | 17
Region of Enrollment [Number; unit: participants]
  United States | 6 | 13 | 19
Histology [Count of Participants; unit: Participants] — In conventional chondrosarcoma, the tumor cells in Grade 1 chondrosarcomas are defined as low-grade, slow-growing tumors with very low metastatic potential. Grade 2 chondrosarcomas are defined as intermediate-grade malignant tumors with the potential to metastasize. Grade 3 chondrosarcomas are highly aggressive with tumor cells actively dividing.
  Participants
    Grade 1 | 2 | 3 | 5
    Grade ≥ 2 | 4 | 9 | 13
    Unknown | 0 | 1 | 1
IDH mutation status [Count of Participants; unit: Participants] — IDH (Isocitrate Dehydrogenase) mutational status was based on available mutational testing obtained by the treating physician prior to study entry.
  Participants
    IDH mutation presence | 2 | 6 | 8
    IDH mutation absence | 4 | 5 | 9
    Unknown | 0 | 2 | 2
Prior lines of treatment [Count of Participants; unit: Participants]
  0 prior lines | 1 | 9 | 10
  1 prior line | 1 | 3 | 4
  2 prior lines | 2 | 1 | 3
  3+ prior lines | 2 | 0 | 2
Prior therapies (by class) [Number; unit: participants] — Per protocol, patients may have been treated with any number of prior systemic therapies. Therefore, one patient may be represented in more than one prior therapy category.
  participants
    Pazopanib | 3 | 1 | 4
    Ivosidenib | 2 | 1 | 3
    Anti-PD1 monotherapy | 2 | 1 | 3
    INBRX-109 | 0 | 1 | 1
    Everolimus | 1 | 0 | 1
    Olutasidenib | 1 | 1 | 2
    Regorafenib | 1 | 0 | 1
    Cabozantinib, Ipilimumab, Nivolumab | 1 | 0 | 1
    Other | 1 | 0 | 1
Prior surgery [Count of Participants; unit: Participants] — Measurement of study participants who had surgery for their metastatic chondrosarcoma prior to beginning study therapy.
  Participants | 5 | 12 | 17
Prior radiation [Count of Participants; unit: Participants] — Measurement of study participants who had radiation to their metastatic chondrosarcoma prior to beginning study therapy.
  Participants | 1 | 5 | 6

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) in Belinostat, ASTX727
Description: Best Objective Response per RECIST Version 1.1 criteria. CR, complete response defined by the disappearance of all target lesions; PR, partial response defined by at least a 30% decrease in the sum of the diameters of target lesions; SD, stable disease defined by neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease; PD, progressive disease defined by at least a 20% increase in the sum of the diameters of target lesions or the appearance of one or more new lesions.
Time Frame: Within 6 months after initiating study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Belinostat, ASTX727)
Number analyzed (Participants) | 13
Participants
  CR/PR | 0
  SD | 6
  PD | 4
  Not Evaluable | 3

2. Secondary Outcome: Presence of Treatment Related Adverse Events (AEs) in Belinostat, ASTX727
Description: Adverse events (AEs) in belinostat, ASTX727 were recorded at each clinical visit and were categorized according to National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. The attribution of AEs to each of the study drugs was recorded and categorized as possibly, probably, or definitely related to treatment. AEs are reported as counts and percentages per AE by grade and the number of patients with a given maximal grade of toxicity.
Time Frame: Up to 24 months post treatment
Population: Treatment-Related Adverse Events Occurring in > 20% of patients treated with belinostat, ASTX727
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Belinostat, ASTX727)
Number analyzed (Participants) | 13
Participants
  Nausea (Grades 1-2) | 9
  Leukopenia (Grades 1-2) | 5
  Leukopenia (Grades 3-4) | 3
  Neutropenia (Grades 1-2) | 1
  Neutropenia (Grades 3-4) | 6
  Anemia (Grades 1-2) | 5
  Anemia (Grades 3-4) | 1
  Fatigue (Grades 1-2) | 5
  Fatigue (Grades 3-4) | 1
  Thrombocytopenia (Grades 1-2) | 4
  Thrombocytopenia (Grades 3-4) | 1
  Infusion Reaction (Grades 1-2) | 4
  Vomiting (Grades 1-2) | 4
  Constipation (Grades 1-2) | 3
  Lymphopenia (Grades 1-2) | 1
  Lymphopenia (Grades 3-4) | 2

3. Secondary Outcome: Progression Free Survival (PFS) in Belinostat, ASTX727
Description: PFS is defined as the time from first treatment with the study drug to the earliest of either disease progression or death from any cause. Patients who are alive and progression free will be censored at the time of their last follow-up. The Kaplan-Meier method was used to evaluate time to event endpoints. Median PFS was reported with a 95% confidence interval. Data will be presented as Kaplan Meier plots.
Time Frame: Time from first treatment with the study drug to the earliest of either disease progression or death from any cause, assessed up to 24 months.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Belinostat, ASTX727)
Number analyzed (Participants) | 13
months | 3.72 [1.83 to NA] — The upper bound Confidence Interval cannot be assessed as there are too few progression events.

4. Secondary Outcome: Presence of Treatment Related Adverse Events (AEs) in Belinostat, SGI-110
Description: Adverse events (AEs) from belinostat, SGI-110 were recorded at each clinical visit and were categorized according to National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. The attribution of AEs to each of the study drugs was recorded and categorized as possibly, probably, or definitely related to treatment. AEs are reported as counts and percentages per AE by grade and the number of patients with a given maximal grade of toxicity.
Time Frame: Up to 24 months post treatment
Population: Treatment-Related Adverse Events Occurring in > 20% of patients treated with belinostat, SGI-110
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Belinostat, SGI-110)
Number analyzed (Participants) | 6
Participants
  Nausea (Grades 1-2) | 4
  Fatigue (Grades 1-2) | 3
  Infusion reaction (Grades 1-2) | 3
  Injection reaction (Grades 1-2) | 3
  Vomiting (Grades 1-2) | 3
  Neutropenia (Grades 1-2) | 1
  Neutropenia (Grades 3-4) | 1
  Pain (Grades 1-2) | 2

5. Secondary Outcome: Progression Free Survival (PFS) in Belinostat, SGI-110
Description: as for outcome 3
Time Frame: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Belinostat, SGI-110)
Number analyzed (Participants) | 6
months | 3.73 [1.87 to NA] — The upper bound Confidence Interval cannot be assessed as there are too few progression events.

6. Secondary Outcome: Objective Response Rate (ORR) in Belinostat, SGI-110
Description: as for outcome 1
Time Frame: Within 6 months after initiating study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Belinostat, SGI-110)
Number analyzed (Participants) | 6
Participants
  CR/PR | 0
  SD | 6
  PD | 0
  Not evaluable | 0

7. Other Pre Specified Outcome: IDH1/2 Mutational Status
Description: Will compare the difference in the objective response rate among patients with IDH1/2 mutations as compared those without IDH1/2 mutations using Fisher's exact test.
Time Frame: Up to 24 months post treatment
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Changes in Expression of Conventional Chondrosarcoma Genes
Description: Data from ribonucleic acid sequencing will be analyzed. Differential expression profiles between baseline and on-treatment samples will be analyzed at the gene level and gene expression changes defined as significant based on absolute log2 fold changes > 2 and adjusted p values < 0.005 for each comparison with consideration of the false discovery rate.
Time Frame: Baseline up to 24 months post treatment
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Changes in Global Deoxyribonucleic Acid Methylation
Description: A Wilcoxon signed-rank test with continuity correction will be used to calculate P values for comparing methylation level distribution at the different time points.
Time Frame: Baseline up to 24 months post treatment
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Changes in Tumor Microenvironment
Description: For quantitative immune multiplexing, data is derived from inForm software, and changes in defined immune cell subsets and expression between baseline and on-treatment samples will be assessed using paired T-tests.
Time Frame: Baseline up to 24 months post treatment
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 24 months post treatment
Description: Adverse events were recorded at each clinical visit and were categorized according to National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. AEs will be reported as counts and percentages per AE by grade and the number of patients with a given maximal grade of toxicity.
Arm/Group | Treatment (Belinostat, SGI-110) | Treatment (Belinostat, ASTX727)
All-Cause Mortality (participants affected / at risk) | 3/6 | 6/13
Serious Adverse Events (participants affected / at risk) | 0/6 | 6/13
Other Adverse Events (participants affected / at risk) | 6/6 | 12/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Belinostat, SGI-110) (N=6) | Treatment (Belinostat, ASTX727) (N=13)
Anemia (Blood and lymphatic system disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Lung infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 2
White blood cell decreased (Investigations) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Concentration Impairment (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Belinostat, SGI-110) (N=6) | Treatment (Belinostat, ASTX727) (N=13)
Anemia (Blood and lymphatic system disorders) | 1 | 6
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 1
Electrocardiogram QT corrected interval prolonged (Cardiac disorders) | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 3
Diarrhea (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 2
Mucositis oral (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 4 | 9
Vomiting (Gastrointestinal disorders) | 3 | 4
Chills (General disorders) | 0 | 1
Fatigue (General disorders) | 3 | 6
Fever (General disorders) | 1 | 0
Infusion related reaction (General disorders) | 3 | 4
Infusion site extravasation (General disorders) | 0 | 1
Injection site reaction (General disorders) | 3 | 1
Pain (General disorders) | 2 | 0
Phlebitis infective (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 0 | 1
Thrush (Infections and infestations) | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 1
CD4 lymphocytes decreased (Investigations) | 0 | 1
Creatinine increased (Investigations) | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 3
Neutrophil count decreased (Investigations) | 2 | 7
Platelet count decreased (Investigations) | 0 | 5
Weight loss (Investigations) | 0 | 1
White blood cell decreased (Investigations) | 1 | 8
Anorexia (Metabolism and nutrition disorders) | 0 | 2
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0
Concentration impairment (Nervous system disorders) | 1 | 1
Dizziness (Nervous system disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Tracheal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Non-pruritic rash (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1
Skin pain (Skin and subcutaneous tissue disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
Phlebitis (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2025-03-25): https://cdn.clinicaltrials.gov/large-docs/43/NCT04340843/Prot_SAP_000.pdf
  • Informed Consent Form: P10330_A09Consent(Redacted).pdf (2025-03-25): https://cdn.clinicaltrials.gov/large-docs/43/NCT04340843/ICF_001.pdf
  • Informed Consent Form: P10330_A09SGIConsent(Redacted).pdf (2025-03-25): https://cdn.clinicaltrials.gov/large-docs/43/NCT04340843/ICF_002.pdf